CLINICAL TRIAL: NCT05937841
Title: Sensitivity of Angiotensin II Type II Receptors in Women Following Preeclampsia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202303202
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Preeclampsia Postpartum
MeSH Terms: interventions — compound 21

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of microvascular function (Experimental): The investigators use intradermal microdialysis to deliver compound 21 and L-NAME to the cutaneous microvasculature
  Interventions: Drug: Compound 21

INTERVENTIONS:
Drug: Compound 21 — AT2R sensitivity: compound 21, and compound 21+ L-NAME (nitric oxide synthase inhibitor) are locally and acutely delivered to the cutaneous microvasculature to assess AT2R-mediated dilation and role of nitric oxide in this response
  Local heating: compound 21 is locally and acutely delivered to the cutaneous microvasculature during local heating of the skin to assess endothelium-dependent dilation, L-NAME is added to assess nitric oxide-dependent dilation during this response

SUMMARY:
Women who develop preeclampsia during pregnancy are more likely to develop and die of cardiovascular disease later in life, even if they are otherwise healthy. The reason why this occurs is unclear but may be related to impaired endothelial function and dysregulation of the angiotensin system that occurs during the preeclamptic pregnancy and persists postpartum, despite the remission of clinical symptoms. The purpose of this investigation is to determine the mechanisms contributing to this lasting blood vessel damage caused by reduced endothelial function in women who have had preeclampsia compared to women who had a healthy pregnancy. Identification of these mechanisms and treatment strategies may lead to better clinical management of cardiovascular disease risk in these women.

The purpose of this study is to examine the microvascular differences in women who have had preeclampsia following activation of protective angiotensin receptors in the skin. This will help increase understanding of the mechanisms of angiotensin II receptors in these women, and how activation of these receptors may restore microvascular function.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) the investigators examine the blood vessels in a dime-sized area of the skin.

ELIGIBILITY:
Inclusion Criteria:

* women who had preeclampsia and women who did not have preeclampsia
* 12 weeks to 5 years postpartum
* 18-45 years old

Exclusion Criteria:

* history of hypertension or metabolic disease before pregnancy
* history of gestational diabetes
* skin diseases
* current tobacco use
* current antihypertensive medication
* statin or other cholesterol-lowering medication
* currently pregnant or planning to become pregnant
* body mass index less than 18.5 kg/m2
* allergy to materials used during the experiment.(e.g. latex),
* known allergy to study drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular blood flow response to local compound 21 treatment measured by laser-Doppler flowmetry | post 1 hour of skin perfusion
  Cutaneous vascular vasodilator response (cutaneous conductance; %max) to exogenous compound 21 perfusion; intradermal microdialysis for the local delivery of compound 21
Change in microvascular endothelial function following local C21 treatment compared to placebo treatment measured by laser-Doppler flowmetry | post 1 hour of skin perfusion
  Cutaneous vascular vasodilator response (cutaneous conductance; %max) to local heating of the skin; intradermal microdialysis for the local delivery of compound 21 compared to control (Ringer's solution), followed by L-NAME infusion to quantify NO-dependent response

SECONDARY OUTCOMES:
Angiotensin receptor expression in endothelial cells | a total of 1 time during the study, within ~4 weeks following enrollment
  Quantify expression of angiotensin II receptor expression in biopsied endothelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Anna Reid-Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz KS, Sun M, Jalal DI, Santillan MK, Stanhewicz AE. Reduced AT2R Signaling Contributes to Endothelial Dysfunction After Preeclampsia. Hypertension. 2025 May;82(5):904-913. doi: 10.1161/HYPERTENSIONAHA.124.24098. Epub 2024 Dec 26. PMID 39723536